CLINICAL TRIAL: NCT07098195
Title: An OPen-label, Multicentre, Single Arm, Clinical InvestigatIon to Evaluate PerFormance and Safety of RIsoR Crest EveRolimus Eluting Coronary Stent System
Brief Title: To Evaluate the Performance and Safety of RisoR Crest Everolimus Eluting Coronary Stent System
Acronym: PACIFIER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poly Medicure Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPL/REG/2025/02
Record Dates: First submitted 2025-07-12; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Percutaneous Coronary Intervention; de Novo Lesions in Native Coronary Arteries
Keywords: RisoR Crest; Everolimus Eluting Stent; Poly Medicure Private Limited; Drug Eluting Stent; Biodegradable Polymer; Pacifier
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: Post-market study in India and Pre-market study in Europe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- RisoR Crest Everolimus Eluting Coronary Stent System (Other): The RisoR Crest Everolimus Eluting Coronary Stent System is coated with a drug and biodegradable polymer coating formulation consisting of Everolimus drug, the active ingredient, and biodegradable polymers.
  This is intended to supply continuous release of Everolimus drug after stent implantation over an extended period of time. The unique ultrasonic atomization drug technology is combined with acoustic activation and carrier stream technologies.
  Interventions: Device: Coronary Stent

INTERVENTIONS:
Device: Coronary Stent — RisoR Crest Everolimus Eluting Coronary Stent System

SUMMARY:
The study will evaluate the performance and safety of RisoR Crest Everolimus Eluting Coronary Stent System. A total of 2000 participants will be included in the study from India and Italy.

DETAILED DESCRIPTION:
The clinical study to evaluate safety and performance of RisoR Crest Everolimus Eluting Coronary Stent System in Coronary Artery Stenosis in Indian (post market) and European (pre-market) Population. Enrolment of up to 1960 participants (100 QCA+50 OCT) in India and 40 in Europe is planned in the current study.

The Primary objective of the study is to evaluate the safety and performance of RisoR Crest Everolimus Eluting Coronary Stent System at 360 days follow up indicated by the Target Lesion Failure (TLF) defined as a hierarchical composite of Cardiac Death, Target Vessel oriented Myocardial Infarction (TV-MI) and Clinically indicated Target Lesion Revascularization (Ci-TLR) at 360 days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System.

The secondary objectives are-

1. To estimate incidence of Device Oriented composite end point (DoCE) which is equivalent of Target Lesion Failure (TLF), a hierarchical composite of Cardiovascular Death, Target Vessel Myocardial Infarction (TV-MI) and Clinically indicated Target Lesion Revascularization (Ci-TLR) at 30, 180 and 270 days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System;
2. Patient oriented composite end point (PoCE), which is a hierarchical composite of any death, any myocardial infarction, any stroke and any coronary revascularization at 30-, 180-, 270- and 360-days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System.
3. Major Adverse Cardiac Events (MACE), a hierarchical composite of cardiovascular death, Myocardial Infarction (MI) and Target Vessel Revascularization (TVR) at 30-, 180-, 270- and 360-days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System.
4. Target Vessel Failure (TVF), a hierarchical composite of cardiovascular death, Target Vessel related Myocardial Infarction (TVMI) and Clinically indicated Target Vessel Revascularization (Ci-TVR) at 30-, 180-, 270- and 360-days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System.
5. Stent thrombosis by ARC 2 and Latency Definitions at 30-, 180-, 270- and 360-days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System and
6. To estimate

   1. Device success, defined as achievement of a final residual diameter stenosis of ≤ 20% (site - reported), using the assigned device only, with Successful deployment of stent and complete retrieval of delivery system without coronary dissection, device disintegration, visible stent malapposition.
   2. procedure success, defined as achievement of a final diameter stenosis ≤ 20%(site-reported) using any PCI method, without the occurrence of death, MI, or repeat target vessel revascularization during hospital stay.
7. To estimate angiographic parameters of performance of RisoR Crest Everolimus Eluting Coronary Stent System as defined by Late Lumen Loss and percentage Diameter Stenosis at 270 days.
8. To estimate percentage of cover struts by OCT at 270 days.

All participants will be followed up at 30±8 days, 180±8 days, 270±10 days and 360±14 days.

For QCA and and OCT sub sets (only for India) all participants will have a mandatory clinic visit at 9 months (270±10 days) for a check angiography and OCT procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years
2. All Genders (Males, Females, Transgenders, Non binary)
3. Patient or legally authorized representative (LAR) agrees to participate by signing the informed consent form.
4. Patient with coronary artery disease eligible for percutaneous coronary intervention (PCI) as per regional or hospital's standard practices guidelines for PCI (For Europe, as per ESC guidelines)
5. Patient with coronary artery disease having one or more de novo or in - stent stenosis lesions in native coronary artery with a visually estimated diameter stenosis ≥70%.
6. Patients with Reference vessel diameter of 2.0 to 4.5 mm
7. Patients with lesion length less than 48 mm

Exclusion Criteria:

1. Pregnant and lactating females
2. Candidates for emergency bypass Surgery
3. Patients corresponding to the criteria of a vulnerable population (Vulnerable subjects, including patients who are unable to fully understand all aspects of the investigation, patients who could be manipulated or unduly influenced, patients lacking capacity in the informed consent procedure and patients with dementia and cognitive impairment, patients under social security, imprisonment etc.)
4. Known congestive heart failure (NYHA IV) or left ventricular ejection fraction (LVEF) less than 30 Percent
5. Patients with known hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, Everolimus or similar drugs, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media
6. Current medical condition with a life expectancy of less than 12 months
7. Patient who have current unstable arrhythmias
8. Patient previously undergone CABG.
9. Left Main Coronary Artery lesion
10. Patients with Cardiogenic shock, systemic bleeding and coagulation disorders, intracranial bleeding, Renal insufficiency requiring dialysis, Acute or chronic renal dysfunction (serum creatinine >2.0mg/dl or 150 μmol/L), peripheral vascular diseases, cancer, etc. and patients who are planning to undergo surgery within 360 days of the index procedure
11. Patients with platelet count <100,000 cells/mm3 or >700,000 cells/mm3 or a WBC <3,000 cells/mm3

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2027-08-17 (Estimated); Study Completion 2028-01-17 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 360 Days
  Target Lesion Failure (TLF) defined as a hierarchical composite of Cardiac Death, Target Vessel oriented Myocardial Infarction (TV-MI) and Clinically indicated Target Lesion Revascularization (Ci-TLR) at 360 days following implantation of RisoR Crest Everolimus Eluting Coronary Stent System.

SECONDARY OUTCOMES:
Incidence of TLF (Equivalent of DoCE) | 30, 180 and 270 days
  1. Cardiovascular Death
  2. Target vessel Myocardial Infarction (TV-MI) and
  3. Clinically indicated Target Lesion Revascularization (Ci-TLR).
Incidence of POCE | 30, 180, 270 and 360 days
  1. All cause death
  2. Any stroke
  3. Any myocardial infarction (includes non-target vessel territory)
  4. Any revascularization
Incidence of MACE | 30, 180, 270 and 360 days
  1. Cardiovascular death
  2. Myocardial Infarction (MI)
  3. Target Vessel Revascularization (TVR)
Target Vessel Failure (TVF) | 30, 180, 270 and 360 days
  Target Vessel Failure (TVF)
Non -Target Vessel related Myocardial Infarction | 30, 180, 270 and 360 days
  Non -Target Vessel related Myocardial Infarction
Stent thrombosis | a. Academic Research Consortium [ARC] 2 definitions - Definite/probable b. As per latency - Acute (0-24 hours), Subacute (24 hours- 30 days) and late (30-360 days)
  Stent thrombosis as per
Device success | Day 0
  defined as achievement of a final residual diameter stenosis of ≤ 20% (site - reported), using the assigned device only, with Successful deployment of stent and complete retrieval of delivery system without coronary dissection, device disintegration, visible stent malapposition
Procedural success | Day 3
  defined as achievement of a final diameter stenosis ≤ 20%(site-reported) using any PCI method, without the occurrence of death, MI, or repeat target vessel revascularization during hospital stay

OTHER OUTCOMES:
QCA Endpoints | 270 days
  In-stent and in-segment % diameter stenosis (DS)
QCA Endpoints | 270 days
  Minimum Lumen Diameter (MLD)
QCA Endpoints | 270 Days
  Late Lumen Loss
QCA Endpoints | 270 Days
  Angiographic binary restenosis
OCT Endpoints | 270 Days
  Diameter Stenosis %
OCT Endpoints | 270 Days
  Proportions of in-stent and in-segment binary restenosis
OCT Endpoints | 270 Days
  Proportion of Struts uncovered and malapposed
OCT Endpoints | 270 Days
  Area restenosis
OCT Endpoints | 270 Days
  Neo-intimal hyperplasia

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Praveen Chandra, DM Cardiology, Principal Investigator — Medanta-The Medicity, Gurugram, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SWL, Tam FCC, Lam SCC, Kong SL, Shea CP, Chan KKW, Wong MKL, Chan MPH, Wong AYT, Yung ASY, Lam YM, Zhang LW, Wu KKY, Mintz GS, Maehara A. The OCT-ORION Study: A Randomized Optical Coherence Tomography Study Comparing Resolute Integrity to Biomatrix Drug-Eluting Stent on the Degree of Early Stent Healing and Late Lumen Loss. Circ Cardiovasc Interv. 2018 Apr;11(4):e006034. doi: 10.1161/CIRCINTERVENTIONS.117.006034. PMID 29654119
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Mahmud E, Pourdjabbar A, Ang L, Behnamfar O, Patel MP, Reeves RR. Robotic technology in interventional cardiology: Current status and future perspectives. Catheter Cardiovasc Interv. 2017 Nov 15;90(6):956-962. doi: 10.1002/ccd.27209. Epub 2017 Aug 10. PMID 28795481
- [Background] Stefanini GG, Holmes DR Jr. Drug-eluting coronary-artery stents. N Engl J Med. 2013 Jan 17;368(3):254-65. doi: 10.1056/NEJMra1210816. No abstract available. PMID 23323902
- [Background] Prati F, Uemura S, Souteyrand G, Virmani R, Motreff P, Di Vito L, Biondi-Zoccai G, Halperin J, Fuster V, Ozaki Y, Narula J. OCT-based diagnosis and management of STEMI associated with intact fibrous cap. JACC Cardiovasc Imaging. 2013 Mar;6(3):283-7. doi: 10.1016/j.jcmg.2012.12.007. PMID 23473109
- [Background] Bangalore S, Amoroso N, Fusaro M, Kumar S, Feit F. Outcomes with various drug-eluting or bare metal stents in patients with ST-segment-elevation myocardial infarction: a mixed treatment comparison analysis of trial level data from 34 068 patient-years of follow-up from randomized trials. Circ Cardiovasc Interv. 2013 Aug;6(4):378-90. doi: 10.1161/CIRCINTERVENTIONS.113.000415. Epub 2013 Aug 6. PMID 23922145
- [Background] Palmerini T, Biondi-Zoccai G, Della Riva D, Mariani A, Genereux P, Branzi A, Stone GW. Stent thrombosis with drug-eluting stents: is the paradigm shifting? J Am Coll Cardiol. 2013 Nov 19;62(21):1915-1921. doi: 10.1016/j.jacc.2013.08.725. Epub 2013 Sep 11. PMID 24036025
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Mehra A, Mohan B. Value of FFR in clinical practice. Indian Heart J. 2015 Jan-Feb;67(1):77-80. doi: 10.1016/j.ihj.2015.02.025. Epub 2015 Mar 14. PMID 25820058
- [Background] Maron DJ, Hochman JS, Reynolds HR, Bangalore S, O'Brien SM, Boden WE, Chaitman BR, Senior R, Lopez-Sendon J, Alexander KP, Lopes RD, Shaw LJ, Berger JS, Newman JD, Sidhu MS, Goodman SG, Ruzyllo W, Gosselin G, Maggioni AP, White HD, Bhargava B, Min JK, Mancini GBJ, Berman DS, Picard MH, Kwong RY, Ali ZA, Mark DB, Spertus JA, Krishnan MN, Elghamaz A, Moorthy N, Hueb WA, Demkow M, Mavromatis K, Bockeria O, Peteiro J, Miller TD, Szwed H, Doerr R, Keltai M, Selvanayagam JB, Steg PG, Held C, Kohsaka S, Mavromichalis S, Kirby R, Jeffries NO, Harrell FE Jr, Rockhold FW, Broderick S, Ferguson TB Jr, Williams DO, Harrington RA, Stone GW, Rosenberg Y; ISCHEMIA Research Group. Initial Invasive or Conservative Strategy for Stable Coronary Disease. N Engl J Med. 2020 Apr 9;382(15):1395-1407. doi: 10.1056/NEJMoa1915922. Epub 2020 Mar 30. PMID 32227755
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612
- [Background] Mauri L, Orav EJ, Candia SC, Cutlip DE, Kuntz RE. Robustness of late lumen loss in discriminating drug-eluting stents across variable observational and randomized trials. Circulation. 2005 Nov 1;112(18):2833-9. doi: 10.1161/CIRCULATIONAHA105.570093. PMID 16267256
- [Background] Hou XM, Han WZ, Qiu XB, Chen H, Fang WY. Safety and effectiveness of drug-eluting stents in Chinese patients with coronary artery disease with off- and on-label indications: results from a single-centre registry. Heart Asia. 2013 Jan 24;5(1):101-5. doi: 10.1136/heartasia-2013-010316. eCollection 2013. PMID 27326098
- [Background] Rosenbaum M. The role of long term beta-blockade after myocardial infarction: Paper 2. Aust Fam Physician. 1978 Jun;Suppl:34-7. PMID 30442
- [Background] Chong B, Jayabaskaran J, Jauhari SM, Chan SP, Goh R, Kueh MTW, Li H, Chin YH, Kong G, Anand VV, Wang JW, Muthiah M, Jain V, Mehta A, Lim SL, Foo R, Figtree GA, Nicholls SJ, Mamas MA, Januzzi JL, Chew NWS, Richards AM, Chan MY. Global burden of cardiovascular diseases: projections from 2025 to 2050. Eur J Prev Cardiol. 2025 Aug 25;32(11):1001-1015. doi: 10.1093/eurjpc/zwae281. PMID 39270739
- See also: World Heart Report 2023: Confronting the World's Number One Killer. — https://world-heart-federation.org/wp-content/uploads/World-Heart-Report-2023.pdf
- See also: Cardiovascular diseases statistics — https://ec.europa.eu/eurostat/statistics-explained/index.php?title=Cardiovascular_diseases_statistics
- See also: India Coronary Stents Market. Coherent Market Insights — https://www.coherentmarketinsights.com/market-insight/india-coronary-stents-market-3484
- See also: Dual Antiplatelet Therapy for 6 Months vs 12 Months After New-generation Drug-eluting Stent Implantation: Matched Analysis of ESTROFA-DAPT and ESTROFA-2 — https://doi.org/10.1016/j.rec.2015.01.008
- See also: CSI: Cardiology Update 2014 — https://www.jaypeedigital.com/book/9789351526186
- See also: The East-West late lumen loss study: Comparison of angiographic late lumen loss between Eastern and Western drug-eluting stent study cohorts — https://doi.org/10.1016/j.ahj.2018.08.017
- See also: MEDICAL DEVICES RULES, 2017 — https://cdsco.gov.in/opencms/resources/UploadCDSCOWeb/2022/m_device/Medical%20Devices%20Rules,%202017.pdf
- See also: Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017 on medical devices, amending Directive 2001/83/EC, Regulation (EC) No 178/2002 and Regulation (EC) No 1223/2009 and repealing Council Directives 90/385/EEC and 93/42/E — https://eur-lex.europa.eu/eli/reg/2017/745/oj/eng